CLINICAL TRIAL: NCT02191566
Title: A Phase II Study of Adjuvant Chemotherapy of S-1 With Oxaliplatin in Gastric Cancer at Stage IIIB/ IV (AJCC 6th) After D2 Resection
Brief Title: S-1/Oxaliplatin for High Risk Patients Who Underwent Gastrectomy
Acronym: SOHUG
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The patient's study enrollment was too low.
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Dong-Hoe Koo, Division of Hematology/Oncology, Department of Internal Medicine, Sungkyunkwan University School of Medicine, Kangbuk Samsung Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOHUG
Record Dates: First submitted 2014-06-23; First posted 2014-07-16 (Estimated); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Stomach Cancer
Keywords: Stomach Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); titanium silicide; tegafur-gimeracil-oteracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- S-1/Oxaliplatin (Experimental): S-1 80 mg/m²/day from day 1 to day 14, every 21 days, for 12 months; Oxaliplatin 130 mg/m² for day 1, every 21 days, for 6 months
  Interventions: Drug: S-1 (452500ACH); Drug: OXALIPLATIN (205803BIJ)

INTERVENTIONS:
Drug: S-1 (452500ACH) — S-1 80 mg/m²/day from day 1 to day 14, every 21 days, for 12 months
  Other Names: TS-1 (tegafur+gimeracil+oteracil)
Drug: OXALIPLATIN (205803BIJ) — Oxaliplatin 130 mg/m² for day 1, every 21 days, for 6 months
  Other Names: PLEOXTIN (645402430)

SUMMARY:
After curative resection, patients with stage IIIB-IV (M0) gastric cancer were given chemotherapy as follows: S-1 orally at 80 mg/m2 divided in two daily doses for 14 days and oxaliplatin at 130 mg/m2 intravenously over 2 h every 21 days as one cycle. S1 was administered for 16 cycles (12 months) and oxaliplatin for 8 cycles (6 months).

ELIGIBILITY:
Inclusion Criteria:

* Patients who voluntarily provide written informed consent prior to entering into this study
* Newly definitely diagnosed with primary gastric or gastroesophageal junction adenocarcinoma histologically
* Patients who underwent radical resection with wide lymph node dissection
* TNM stage (6th AJCC) of IIIB or IV on post-operative staging
* Patients who can be randomized within 6 weeks after surgery

Exclusion Criteria:

* Aged < 20 years or ≥ 76 years
* Eastern Cooperative Oncology Group (ECOG) performance status >2
* Patients who underwent surgery for neoplasm in stomach in the past
* History of malignant disease The following cases can be included in this study - adequately treated basal cell or squamous cell skin cancer, cervical carcinoma in situ
* Gastric or gastroesophageal junction adenocarcinoma with distant metastasis (M1) including distant lymph node (behind the pancreas, along the aorta, portal vein, behind the peritoneum, mesenteric lymph node)
* Residual cancer on post-operative staging (R1 and R2 resection)
* Patients who received adjuvant chemotherapy, or neoadjuvant chemotherapy and/or radiotherapy and/or immunotherapy in the past for treatment of gastric cancer
* Any of the following within 6 months prior to the study recruitment: Myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass, NYHA class III or IV congestive heart failure, stroke or transient ischemic attack, serious cardiac arrhythmia requiring treatment
* Patients of childbearing potential who do not agree to use generally accepted effective method of birth control during the study treatment period and for at least 6 months after the end of study treatment
* Pregnant women, breastfeeding women, or women of childbearing potential whose pregnancy test result is positive•
* History of hypersensitivity to the investigational products (S1 and Oxaliplatin)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
3-year recurrence-free survival, RFS | 3-year

SECONDARY OUTCOMES:
5-year overall survival, OS | 5-year

OTHER OUTCOMES:
Toxicity will be graded according to the CTCAE. | 1-year
  For patients who have experienced a dosing delay for starting treatment cycle, all assessments will be performed as scheduled. Reasons for dose modifications or delays, the supportive measures taken, and the outcome will be documented in the patient's chart and recorded in the CRF.
compliance for chemotherapy | 1-year
  Accountability and subject compliance will be assessed by maintaining adequate dose of S1 and return records. Subjects will be asked to return all used and unused drug supply containers at the end of each cycle as a measure of compliance. The clinical administration records will be used to monitor compliance with oxaliplatin.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Hoe Koo, MD,PhD, Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

REFERENCES:
- [Background] Sasako M, Sakuramoto S, Katai H, Kinoshita T, Furukawa H, Yamaguchi T, Nashimoto A, Fujii M, Nakajima T, Ohashi Y. Five-year outcomes of a randomized phase III trial comparing adjuvant chemotherapy with S-1 versus surgery alone in stage II or III gastric cancer. J Clin Oncol. 2011 Nov 20;29(33):4387-93. doi: 10.1200/JCO.2011.36.5908. Epub 2011 Oct 17. PMID 22010012
- [Background] Bang YJ, Kim YW, Yang HK, Chung HC, Park YK, Lee KH, Lee KW, Kim YH, Noh SI, Cho JY, Mok YJ, Kim YH, Ji J, Yeh TS, Button P, Sirzen F, Noh SH; CLASSIC trial investigators. Adjuvant capecitabine and oxaliplatin for gastric cancer after D2 gastrectomy (CLASSIC): a phase 3 open-label, randomised controlled trial. Lancet. 2012 Jan 28;379(9813):315-21. doi: 10.1016/S0140-6736(11)61873-4. Epub 2012 Jan 7. PMID 22226517
- [Background] Lee SS, Jeung HC, Chung HC, Noh SH, Hyung WJ, Ahn JY, Rha SY. A pilot study of S-1 plus cisplatin versus 5-fluorouracil plus cisplatin for postoperative chemotherapy in histological stage IIIB-IV (M0) gastric cancer. Invest New Drugs. 2012 Feb;30(1):357-63. doi: 10.1007/s10637-010-9515-2. Epub 2010 Aug 24. PMID 20734110